CLINICAL TRIAL: NCT03128476
Title: Effects of the Supplementation of Essence of Chicken on Physical Fatigue and Brain Functions Such as Working Memory and Attention Among Healthy Adults
Brief Title: Effects of Essence of Chicken on Physical Fatigue, Working Memory and Attention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sprim Advanced Life Sciences (Other)
Collaborators: Cerebos (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BEC
Record Dates: First submitted 2017-02-20; First posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-02

CONDITIONS: Healthy Subjects; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 bottle (Active Comparator)
  Interventions: Dietary Supplement: Essence of Chicken
- 2 bottles (Active Comparator)
  Interventions: Dietary Supplement: Essence of Chicken
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo (Energy matched)

INTERVENTIONS:
Dietary Supplement: Essence of Chicken — Brand's Essence of Chicken (BEC) is produced via a water extraction process from chicken meat for several hours under high-temperature, followed by centrifugation to remove fat and cholesterol, vacuum concentration to 3- to 4-fold, sterilization by high temperature and pressure before bottling. This kind of chicken essence is rich in protein, and low in sugar and fat, conveniently available and consumable, and easy for household storage.
  Arms: 1 bottle; 2 bottles
Dietary Supplement: Placebo (Energy matched)
  Arms: Placebo

SUMMARY:
In Southeast Asia, Essence of Chicken, a chicken-meat-extract, is a popular beverage and is consumed as a traditional remedy for several ailments, including the use as a nutritional supplement for sickness, enhancement of mental efficiency, and recovery from mental fatigue. While the elderly use it as a nutritional supplement, students use it for relief from anxiety during exam times.

The present study is conducted in order to assess the effects of BEC on various physical and mental parameters including physical fatigue, working memory and attention, mood and stress, in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Normal BMI
* Not continuously taken Essence of Chicken for the last 3 months
* Physical and psychological fatigue inclusion criteria/test/cutoff using CFQ (where individuals' CFQ scores 4 or above)

Exclusion Criteria:

* Suffering from chronic or malignant diseases e.g. cancer, heart, liver, renal or other metabolic diseases.
* Any psychiatric or neurological disease
* Pregnant and lactating women
* Subjects participated in any investigational drug trial within 4 weeks before screening
* Consumption of food supplement in the previous 2 weeks
* Professional athletes
* Subjects with recent lifestyle changes in the past 4 weeks
* History of allergy to chicken meat and seafood

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 364 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2016-11-07 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Fatigue-vitality | 4 weeks
  Psychometric tests SF-36 (score 100%)
Physical fatigue | 4 weeks
  Chalder Fatigue Questionnaire (score 0-33)
Attention | 4 weeks
  Stroop (mean latency and proportion correct)
Sustained attention | 4 weeks
  Sustained Attention to Response Task (mean latency and % of correct trials)
Working memory | 4 weeks
  Digit Span test (Maximal FORWARD digit span and Maximal BACKWARD digit span, etc)

SECONDARY OUTCOMES:
Mood | 4 weeks
  POMS brief is used as a psychometric test to measure mood (6 domains).
Stress | 4 weeks
  DASS is used as a psychometric test to measure stress (score 0-42).
Adverse effects | 4 weeks
  Comparison of adverse events on IP and placebo groups.